CLINICAL TRIAL: NCT00452751
Title: Multi-institutional Prospective Randomized Trial on the Assessment of Laparoscopic Surgery for Gastric Cancer
Brief Title: Comparison of Laparoscopic Versus Open Gastrectomy for Gastric Cancer: A Prospective Randomized Trial
Acronym: KLASS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0520310-2
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; laparoscopic surgery; survival; preoperative staging; morbidity; quality of life; acute inflammatory reaction; cost
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: laparoscopy-assisted distal gastrectomy
Procedure: open distal gastrectomy

SUMMARY:
The purpose of this study is to assess the usefulness of laparoscopic surgery for gastric cancer in comparison with open gastrectomy.

DETAILED DESCRIPTION:
Recently, in technical aspects, almost all kinds of open gastric cancer surgeries can be reproduced laparoscopically. However, many controversies exist due to no evidence and no long-term results. There was no prospective multi-center large-scale randomized controlled trial in the world on the long-term outcome of laparoscopic gastric cancer surgery.

Korean Laparoscopic Gastrointestinal Surgery Study Group, therefore, proposed a multi-institutional prospective randomized trial on comparing laparoscopy-assisted versus open distal gastrectomy for gastric cancer (KLASS Trial) after the feasibility and validity of these procedures had been evaluated by analyzing retrospective multi-center large series.

This KLASS trial is supported by a grant for 2005 from the National R&D Program for Cancer Control, Ministry of Health & Welfare, Republic of Korea. Nine surgeons from 9 centers are participating in this trial. All the participants performed more than 50 cases of open and laparoscopic gastrectomies, respectively and their institutes had more than 80 cases of gastric cancer surgeries per year. Primary endpoint of this trial is to elucidate that there is no difference of overall and disease-free survivals between laparoscopic and open groups. The KLASS trial consists of 5 major subjects: comparison of 5-year overall and disease-free survivals, standardization of preoperative diagnosis, assessment of the quality of life, evaluation of postoperative inflammatory response and immune function, and cost-effectiveness. The KLASS trial will be able to validate and verify laparoscopic gastric cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically proven gastric adenocarcinoma
2. age: 20 ~ 80 years
3. preoperative stage: cT1N0M0, cT1N1M0, cT2aN0M0
4. no history of other cancer
5. no history of chemotherapy or radiotherapy
6. written informed consent

Exclusion Criteria:

1. ASA >3
2. combined resection
3. total gastrectomy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2006-02; Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
overall survival

SECONDARY OUTCOMES:
disease-free survival
morbidity and mortality
quality of life
inflammatory and immune response
cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Hyung-Ho Kim, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital, 300 Gumi-dong, Bundang-gu, Seongnam-si, Gyeonggi-do, 463-707, Korea
Locations (16):
- South Korea (16):
  - Chungnam National University Hospital, Daejun, Chungcheongnam-do
  - Chonbuk National University Hospital, Chonjoo, Jeollabuk-do
  - Soonchunhyang University College of Medicine, Bucheon-si
  - Catholic University Holy Family Hospital, Bucheon-si
  - Keimyung University College of Medicine, Daegu
  - Dong-A University College of Medicine, Pusan
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Yonsei University College of Medicine, Seoul
  - Catholic University Kangnam St. Mary's Hospital, Seoul
  - Ewha Womans University Hospital, Seoul
  - Kangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Ajou University College of Medicine, Suwon
  - St. Vincent's Hospital, Suwon
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Derived] Kim HH, Han SU, Kim MC, Kim W, Lee HJ, Ryu SW, Cho GS, Kim CY, Yang HK, Park DJ, Song KY, Lee SI, Ryu SY, Lee JH, Hyung WJ; Korean Laparoendoscopic Gastrointestinal Surgery Study (KLASS) Group. Effect of Laparoscopic Distal Gastrectomy vs Open Distal Gastrectomy on Long-term Survival Among Patients With Stage I Gastric Cancer: The KLASS-01 Randomized Clinical Trial. JAMA Oncol. 2019 Apr 1;5(4):506-513. doi: 10.1001/jamaoncol.2018.6727. PMID 30730546
- [Derived] Kim W, Kim HH, Han SU, Kim MC, Hyung WJ, Ryu SW, Cho GS, Kim CY, Yang HK, Park DJ, Song KY, Lee SI, Ryu SY, Lee JH, Lee HJ; Korean Laparo-endoscopic Gastrointestinal Surgery Study (KLASS) Group. Decreased Morbidity of Laparoscopic Distal Gastrectomy Compared With Open Distal Gastrectomy for Stage I Gastric Cancer: Short-term Outcomes From a Multicenter Randomized Controlled Trial (KLASS-01). Ann Surg. 2016 Jan;263(1):28-35. doi: 10.1097/SLA.0000000000001346. PMID 26352529
- [Derived] Kim HH, Han SU, Kim MC, Hyung WJ, Kim W, Lee HJ, Ryu SW, Cho GS, Kim CY, Yang HK, Park DJ, Song KY, Lee SI, Ryu SY, Lee JH; Korean Laparoscopic Gastrointestinal Surgery Study (KLASS) Group. Prospective randomized controlled trial (phase III) to comparing laparoscopic distal gastrectomy with open distal gastrectomy for gastric adenocarcinoma (KLASS 01). J Korean Surg Soc. 2013 Feb;84(2):123-30. doi: 10.4174/jkss.2013.84.2.123. Epub 2013 Jan 29. PMID 23396494
- [Derived] Kim HH, Hyung WJ, Cho GS, Kim MC, Han SU, Kim W, Ryu SW, Lee HJ, Song KY. Morbidity and mortality of laparoscopic gastrectomy versus open gastrectomy for gastric cancer: an interim report--a phase III multicenter, prospective, randomized Trial (KLASS Trial). Ann Surg. 2010 Mar;251(3):417-20. doi: 10.1097/SLA.0b013e3181cc8f6b. PMID 20160637
- [Derived] Kim MC, Kim W, Kim HH, Ryu SW, Ryu SY, Song KY, Lee HJ, Cho GS, Han SU, Hyung WJ; Korean Laparoscopic Gastrointestinal Surgery Study (KLASS) Group. Risk factors associated with complication following laparoscopy-assisted gastrectomy for gastric cancer: a large-scale korean multicenter study. Ann Surg Oncol. 2008 Oct;15(10):2692-700. doi: 10.1245/s10434-008-0075-z. Epub 2008 Jul 29. PMID 18663532